CLINICAL TRIAL: NCT02978560
Title: Indocyanine Green Tissue Perfusion Monitoring
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Baltimore Medical & Surgical Associates PA (Unknown)
Responsible Party: Principal Investigator, Stephen R Thom, Professor, University of Maryland, Baltimore
Other Study IDs: HP-00071920
Record Dates: First submitted 2016-11-23; First posted 2016-12-01 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Regional Blood Flow; Wound Heal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- control: The source population for this cohort will be 30 healthy individuals with no know cardiovascular disease or wound healing defects. Subjects will be recruited by word-of-mouth, who receive no remuneration and who will be selected for the study on the basis of inclusion and exclusion criteria. They will undergo fluorescence-mediated photoplethysmography once.
  Interventions: Diagnostic Test: fluorescence-mediated photoplethysmography
- Wound Group: The source population will be 30 patients who present to wound care clinic with Diabetic Foot Ulcers. Candidate subjects will have had a standard wound evaluation and medical history taken as a matter of their standard of care. On the basis of the evaluation, the physician-investigators will determine if the patient meets the eligibility criteria. If so, the study will be explained to the patient at that time, and Informed Consent will be obtained. 30 healthy subjects will also be included, recruited by word-of-mouth, who receive no remuneration and who will be selected for the study on the basis of the following inclusion and exclusion criteria. They will undergo fluorescence-mediated photoplethysmography once at the onset of their wound care.
  Interventions: Diagnostic Test: fluorescence-mediated photoplethysmography

INTERVENTIONS:
Diagnostic Test: fluorescence-mediated photoplethysmography — Indocyanine green dye (ICG) will be injected intravenously as a sterile solution at a dose of 0.5 mg/kg, and then imaging of skin will be done with a fluorescence camera. The ICG-angiogram sequence will consist of 1.5 x 2.0-cm field-of-view ICG fluorescence images acquired at the rate of approximately 30/sec during a period of about 15 seconds. Following acquisition of the initial transit angiogram sequence, several additional 15-second-long image sequences will be acquired during the next half-hour, but without any additional injections.

SUMMARY:
The aim of this project is to demonstrate that fluorescence-mediated photoplethysmography (FM-PPG) is capable of routinely acquiring the tissue perfusion data sufficient to detect and monitor skin tissue perfusion anomalies.

DETAILED DESCRIPTION:
Methods to reliably predict which cutaneous wounds will heal are unreliable and clinical judgment inadequate. This is a problem for all health care providers and a common dilemma when evaluating patients in the Emergency Department. While capillary blood perfusion of the skin is a recognized requirement for healing, objective methods to reliably quantify this necessary physiological parameter are lacking. In large part, this is due to difficulties visualizing and recording capillary blood flow. Despite technical advances in blood flow imaging the capillary circulation remains poorly characterized. That is, current methodology can only image medium-to-large caliber vessels, not the small capillaries. The investigators hypothesize that with new technology, objective assessment of capillary flow can be achieved with fluorescence-mediated photoplethysmography (FM-PPG) methodology, and this evaluation can be used to objectively determine which wounds will heal promptly versus require adjunctive interventions.

FM-PPG is currently being used clinically in clinics worldwide as a way to image blood flow, but the apparatus provides only a relative measurement. Thus, this investigation is Observational in nature and not Interventional. With repeated evaluations over weeks, current FM-PPG allows an assessment to be made on whether wound conditions are improving. The investigators have a device containing new imaging software which, in theory, can offer precise quantification of capillary blood flow. If true, a single measurement may provide the data necessary to predict which patients are in danger of not healing and thus requiring aggressive, and at times expensive or painful interventions and - even worse - limb amputations. This protocol is to test proof-of-concept by first evaluating cutaneous capillary follow in 30 normal, healthy individuals and then 30 individuals presenting for treatment with a variety of skin wounds to a clinic.

FM-PPG methodology requires intravenous injection of a small amount of a fluorescent dye, indocyanine green (ICG). ICG is an FDA-approved agent that has been safely used in over 4000 patients. The area of skin to be measured is positioned below a camera and low-power laser instrument to take fluorescent pictures. The ICG is dissolved in sterile salt water for injection and about one and one half tablespoons injected into a vein. Typically, the measuring sequence consists of obtaining fluorescence images at the rate of approximately 30/second during a period of about 15 seconds. Following acquisition of the initial transit angiogram sequence, several additional 15-second-long image sequences are then acquired during the next half-hour, but without any additional injections. At about 60 seconds following dye injection, about two teaspoons of venous blood is withdrawn. This blood is used in the laboratory to determine the ICG dye concentration as a verification of the concentration determined by the camera images as part of the FM-PPG software algorithm (circulating dye concentration is needed in calculation of quantitative blood perfusion).

Since this study will be the first to employ a methodology capable of acquiring absolute tissue blood perfusion data from multiple subjects, there exists no database to indicate the normal range of variation in skin tissue perfusion that occurs in normal subjects. Since abnormal perfusion cannot be clearly recognized until the normal range of variation has been established, the first 30 subjects will be normal individuals. Then the following 30 subjects will be patients undergoing wound healing therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, of any ethnic background, who are at least 21 years of age and have normal healthy skin (30 normal subjects) or patients with diabetic foot ulcer lesions (30 patients).
2. All subjects must be willing and be able to comply with the protocol, and to provide informed consent.

Exclusion Criteria:

1. Patient currently participating in any other drug or device investigational study.
2. Patient with significant liver or kidney disease.
3. Patient with known adverse reaction to indocyanine green or iodine.
4. Patient is pregnant or nursing.
5. Patient with peripheral vascular disease and an ankle-brachial index blood flow of 0.6 or less

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Indocyanine Green Tissue Perfusion Monitoring | 2 years
  Flow measurements on normal skin and sites of diabetic neuropathic wounds

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Thom, MD, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Baltimore Medical & Surgical Associates PA, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Flower RW, Mirza Z, Thom SR. Absolute quantification (ml blood/sec * mm2 tissue) of normal vs. diabetic foot skin microvascular blood perfusion: Feasibility of FM-PPG measurements under clinical conditions. Microvasc Res. 2019 May;123:58-61. doi: 10.1016/j.mvr.2018.12.004. Epub 2018 Dec 24. PMID 30590061